CLINICAL TRIAL: NCT05020470
Title: Pilot Testing A Theory-Driven Self-Management Intervention for Chronic Musculoskeletal Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00290512
Record Dates: First submitted 2021-08-19; First posted 2021-08-25 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-06

CONDITIONS: Chronic Musculoskeletal Pain
Keywords: Chronic Pain; Musculoskeletal; Auricular Point Acupressure
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Intervention Model Description: This prospective, multisite study will randomly assign at least 30 participants into three groups: (1) Self-guided mAPA (S-mAPA), (2) In-Person Training + mAPA (IP-mAPA), and (3) Usual Care Control (UC). Data will be collected at pre- (T1), post-completion of intervention (T2), follow-ups at post 1M- (primary endpoint) (T3), 2M (T4), and 3M (secondary endpoint, long-term sustained effect) (T5) for a total of four assessments. Participants assigned to IP-mAPA but are unable to come in for the in person training can choose to be in the S-mAPA group; this data will be collected. EMA will be used to assess momentary pain outcomes and APA adherence. This pilot study will collect feasibility and pain-related outcomes at more than 1 study site. The consent process will occur virtually (via secure email). Due to the nature of this pilot study, the anticipated enrollment will be a total of at least N = 30.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Participants cannot be masked to the three treatment groups. The PI and Co-Is will be blinded regarding group assignment and will not contact or interact with the participants during the intervention and outcome assessments. Data collector for outcome assessments will be blinded since there will be no seeds placed on the ears when the data are collected.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Self-guided mAPA (S-mAPA) (Experimental): S-mAPA group will be provided with instructions so that participants can learn to self-administer APA weekly for four weeks and then followed by weekly telecommunication for Q & As.
  Interventions: Device: Virtual Auricular Point Acupressure (APA)
- In-Person Training + mAPA (IP-mAPA) (Experimental): Participants will receive one in-person training after baseline data is collected and then will self-administer APA on the same schedule with weekly telecommunication as those in the mAPA group.
  Interventions: Device: Virtual Auricular Point Acupressure (APA); Other: In-Person Training
- Usual Care Control (UC) (Active Comparator): Participants will receive usual care only for their pain; after enrolled, patients will receive weekly telecommunication to control for attention and time. The content of the phone/video call will focus on the pain problem they have and the investigators will provide additional information published by the National Center for Complementary and Integrative Health "Chronic Pain: In-Depth" (https://www.nccih.nih.gov/health/chronic-pain-in-depth) which the investigators used in the R01 study for participants enrolled in the control group
  Interventions: Other: Usual Care

INTERVENTIONS:
Device: Virtual Auricular Point Acupressure (APA) — Participants will learn how to self-administer APA by themselves.
  Arms: In-Person Training + mAPA (IP-mAPA); Self-guided mAPA (S-mAPA)
Other: In-Person Training — Participants will receive in-person training to self-administer APA.
  Arms: In-Person Training + mAPA (IP-mAPA)
Other: Usual Care — Participants will continue to do whatever they are instructed by theirs physicians.
  Arms: Usual Care Control (UC)

SUMMARY:
The proposed randomized control trial will evaluate auricular point acupressure (APA) treatment administered by the participant themselves with the use of a phone app on chronic musculoskeletal pain (CMP) outcomes.

This study will randomly assign participants into three groups: (1) Self-guided mAPA (S-mAPA), (2) In-Person Training + mAPA (IP-mAPA), and (3) Usual Care Control (UC). EMA will be used to assess momentary pain outcomes and APA adherence.

Data will be collected at pre- (T1), post-completion of intervention (T2), follow-ups at post 1M- (primary endpoint) (T3), 2M (T4), and 3M (secondary endpoint, long-term sustained effect) (T5) for a total of four assessments.

DETAILED DESCRIPTION:
Chronic musculoskeletal pain (CMP) is the most common self-reported and clinically diagnosed pain condition in the US and costs up to $635 billion annually. Analgesics/opioids are the most common treatments utilized by patients with CMP, however, unnecessary opioid use has resulted in the current opioid epidemic. The Institute of Medicine recommended guidelines for non-pharmacologic, self-management strategies to manage pain. However, these guidelines have not been broadly implemented due to time constraints among healthcare providers, accessibility, patient's beliefs/motivations, and high cost/insurance coverage, especially among socioeconomically disadvantaged and vulnerable patients.

Auricular point acupressure (APA), a non-invasive procedure, provides acupuncture-like stimulations on ear points using small pellets instead of needles to self-manage pain. The investigator's interdisciplinary team has accumulated extensive evidence (11 clinical trials) supporting the efficacy of interventionist-administered APA to manage pain. The randomized clinical trial (RCT) comparing APA to sham APA demonstrated: (1) Significant rapid and sustained effect: APA resulted to ≥38% rapid pain relief among participants at three minutes post-APA; >44% pain relief and >28% improved physical function at follow-up after 4-weeks APA; (2) Reduced use of medications: After 4-weeks of APA, ≥60% of participants reported less use of pain medications; and (3) Significant impact on physiological measures: APA controls pain through blocking pro-inflammatory cytokines (IL-1β, IL-2) and modulating nerve sensitivity. No adverse effects from APA were reported.

The investigator's long-term goal is to eliminate pain care disparities and reduce society's reliance on opioids to manage pain. Leveraging technology, the proposed study will help advance mAPA, a novel, easy-to-initiate, rapid, safe, and non-pharmacologic tool incorporated in a self-management plan to manage pain in real-world settings. The proposed intervention promises to provide important and timely information to advance a non-opioid and self-managed pain treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years of age or older.
* Receiving outpatient pain treatment for CMP condition (e.g., pain in the back, hip, knee, upper extremity, lower extremity, neck, pelvic, headache/migraine).
* Chronic pain ≥ 4 on a scale of 0-10 point numerical pain, persisting for at least 3 months or has resulted in pain on at least half the days in the past 6 months.

Exclusion Criteria:

* Disease that might confound therapeutic effects or explanation of outcomes, i.e., infection, malignant tumors, or autoimmune diseases.
* Severe ear skin issues.
* Use of some types of hearing aids (size may obstruct the placement of seeds)
* Concurrent major psychiatric disorder (i.e., participant self-report).
* Pregnant women will be excluded from the study based on the self-reported data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2021-09-22 (Actual); Primary Completion 2022-08-11 (Actual); Study Completion 2022-08-11 (Actual)

PRIMARY OUTCOMES:
Pain intensity | Up to 4 months
  The Brief Pain Inventory-short form (BPI-sf) questionnaire includes assessment of pain location and multiple aspects of severity of pain, numbness, tingling, and stiffness, including worst, least, average pain, and present, as well as the interference with daily activities. The Brief Pain Inventory-short form (BPI-sf) has a total score ranging from 0 to 10 with higher scores indicating more pain.
Pain Interference | Up to 4 months
  The Roland Morris Disability Questionnaire (RMDQ), 24-item measure, was used to assess the impact of back pain on their daily functioning. The score ranged from 0 (no disability) to 24 (maximum disability).
Physical Function | Up to 4 months
  The Oswestry Disability Index (ODI) was used to measure a participants impairment and quality of life on 10 items with 0-5 point scales. Each section is scored on a 0-5 scale, 5 representing the greatest disability. The index is calculated by dividing the summed score by the total possible score, which is then multiplied by 100 and expressed as a percentage. Thus, for every question not answered, the denominator is reduced by 5; a lower score indicates less disability.

SECONDARY OUTCOMES:
Health Related Quality of Life (HRQoL) | Up to 4 months
  The WHO Quality of Life-BREF (WHOQOL-BREF), used to measure quality of life. The WHOQOL-BREF, is self-administered, and measures the following broad domains: physical health, psychological health, social relationships, and environment. Each individual item of the WHOQoL is scored from 1 to 5 on a response scale, which is stipulated as a five-point ordinal scale. The measure is calculated by summing the point values for the questions corresponding to each domain and then transforming the scores to a 0-100 point interval. The first two questions of the WHOQOL-BREF do not correspond to a domain, but are meant to provide a global assessment of quality of life. Higher scores in each of the domains correspond to greater perceived quality of life.
Treatment Satisfaction | Up to 4 months
  The participants will be assessed using a 12-item Treatment Satisfaction Questionnaire, with 4 items with scored for treatment difficulty 1 (extremely difficult) - 5 (not difficult), 7 single-choice questions assessing satisfaction and effectiveness of treatment and 3 open-ended questions assessing satisfaction and effectiveness of treatment. Maximum score of 36; A higher score indicates more satisfaction from the treatment.
Fear-Avoidance | Up to 4 months
  It is measured by Fear-avoidance beliefs questionnaire (FABQ) that focuses on participants beliefs about how physical activity and work affect their pain. The questionnaire consists of 16 items in which a participant rates their agreement with each statement on a 7-point Likert scale. Where 0= completely disagree, 6=completely agree. Maximum score of 96; A higher score indicates more strongly held fear-avoidance beliefs. The first 5 questions pertain to physical activity while the remaining 11 pertain to work. The Physical Activity subscale range 0-24 is the sum of items 2-5; the Work subscale, range 0-42 is the sum of items 6, 7, 9-12 and 15.
Placebo effect | Up to 4 months
  Placebo effects will be measured via Healing Encounters and Attitudes Lists (HEAL) Treatment Expectation questionnaire. HEAL is an item bank comprised of 6 domains. The Treatment Expectancy questionnaire consists of 6 items on a 5 point scale - not at all to very much. Score range of 6-30 with higher score indicating better outcome.
Pain and Catastrophizing Scale (PCS) | Up to 4 months
  The PCS was included to detect exaggerated and negative interpretations of pain. It is a self-report scale that consists of 13 items. Participants were asked to reflect on past painful experiences and to indicate to which degree he/she experienced symptoms such as helplessness or rumination when feeling pain.This is a 0-4 Likert scale (score sum 0-52) with responses ranging from "not at all" to "all the time," and high scores indicate stronger catastrophizing.
Positive Outlook | Baseline and 4 months
  Pre and post treatment positive outlook effects will be measured via Healing Encounters and Attitudes Lists (HEAL) Positive Outlook scale. The participants will be assessed using a 6-item questionnaire, scored for outlook on life 1 (not at all) - 5 (very much). Score range of 6- 30; A higher score indicates more positive outlook and satisfaction with ones life.

CONTACTS AND LOCATIONS:
Overall Officials: Chao Hsing Yeh, PhD, Principal Investigator — Johns Hopkins School of Nursing; Jennifer Kawi, PhD, Principal Investigator — University of Nevada, Las Vegas
Locations (2):
- United States (2):
  - Johns Hopkins School of Nursing, Baltimore, Maryland
  - University of Nevada, Las Vegas, Las Vegas, Nevada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kawi J, Yeh CH, Lukkahatai N, Hardwicke RL, Murphy T, Christo PJ. Exploring the Feasibility of Virtually Delivered Auricular Point Acupressure in Self-Managing Chronic Pain: Qualitative Study. Evid Based Complement Alternat Med. 2022 Aug 29;2022:8079691. doi: 10.1155/2022/8079691. eCollection 2022. PMID 36072397
- [Background] Yeh CH, Kawi J, Ni A, Christo P. Evaluating Auricular Point Acupressure for Chronic Low Back Pain Self-Management Using Technology: A Feasibility Study. Pain Manag Nurs. 2022 Jun;23(3):301-310. doi: 10.1016/j.pmn.2021.11.007. Epub 2021 Dec 25. PMID 34961729
- [Background] Kawi J, Yeh CH, Li M, Caswell Bs K, Mazraani Md M, Lukkahatai PhD Rn N, Mensah Rn S, Taylor J, Budhathoki C, Christo P. Auricular Point Acupressure Smartphone Application to Manage Chronic Musculoskeletal Pain: A Longitudinal, One-Group, Open Pilot Trial. Glob Adv Health Med. 2021 Jan 22;10:2164956120987531. doi: 10.1177/2164956120987531. eCollection 2021. PMID 33623727
- [Result] Yeh CH, Kawi J, Grant L, Huang X, Wu H, Hardwicke RL, Christo PJ. Self-Guided Smartphone Application to Manage Chronic Musculoskeletal Pain: A Randomized, Controlled Pilot Trial. Int J Environ Res Public Health. 2022 Nov 11;19(22):14875. doi: 10.3390/ijerph192214875. PMID 36429591
- [Derived] Kawi J, Yeh CH, Grant L, Huang X, Wu H, Hua C, Christo P. Retention, adherence, and acceptability testing of a digital health intervention in a 3-group randomized controlled trial for chronic musculoskeletal pain. Complement Ther Med. 2024 May;81:103030. doi: 10.1016/j.ctim.2024.103030. Epub 2024 Mar 2. PMID 38437926

DOCUMENTS (1):
  • Informed Consent Form (2021-08-12): https://cdn.clinicaltrials.gov/large-docs/70/NCT05020470/ICF_000.pdf